CLINICAL TRIAL: NCT06106659
Title: Comparison of Clinical Outcomes of Mini Midline Catheters With Different Placement Sites: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Zhao Linfang, Assitant nursing director, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-802-01
Record Dates: First submitted 2023-10-09; First posted 2023-10-30 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Catheter Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- forearm (Experimental): Mini midline catheter forearm placement.
  Interventions: Device: Mini Midline
- upper arm (Other): Mini midline catheter upper arm placement
  Interventions: Device: Mini Midline

INTERVENTIONS:
Device: Mini Midline — The tube was placed in the upper arm in the test group and in the forearm in the control group. The veins were selected according to anatomical criteria (vein diameter and depth), and the puncture site was protected with a sterile cavity towel. The cannulation nurse wore sterile gloves and injected local anesthesia (1 mL of lidocaine) before venipuncture. Venipuncture was always performed using real-time ultrasound-guided visualization of the vein-guiding needle using an "out-of-plane" approach, and once the tip of the needle was visualized within the vein and the blood flowed back through the needle, a guidewire was introduced and the needle was removed. After the needle is removed, the cannula is advanced into the vein, the guidewire is removed, and the cannula is attached to an extension cord closed with a needleless connector.

SUMMARY:
Peripheral venous catheters are the most commonly used vascular access devices in healthcare today, including indwelling needles, mini-midline catheters, and medium-length venous catheters. Peripheral venous catheters are required due to clinical needs for prescribed intravenous treatments, medications, surgical procedures, or diagnostics, such as computed tomography scans, etc. One study noted that more than 70% of hospitalized patients had indwelling needles placed. However, post-placement failure of indwelling needles occurs in 30%-50% of patients before completing treatment, unplanned catheter failure occurs in 69% of patients before completing treatment, and there is a 30%-60% risk of various complications. And patients are often subjected to repeat catheter placement, such as improper catheter placement or improperly entered medications. In addition, catheterization is prone to infectious and noninfectious complications, and the risk of phlebitis increases 4.4-fold when catheters are reintroduced.Tan et al. found that the average number of indwelling needle insertions per patient admission was 2.82, and therefore, approximately 44% of adult patients required more than one indwelling needle to complete IV therapy during their hospitalization. According to Helm et al, multiple insertions of indwelling needles per patient lead to unnecessary pain and anxiety, and multiple attempts per insertion further increase the risk of complications. These also lead to prolonged hospitalization, additional healthcare costs, pain, anxiety, and other adverse experiences.

DETAILED DESCRIPTION:
Therefore, alternative vascular access is needed to meet the needs of patients. The mini midline catheter is a novel vascular access in recent years that is smaller in diameter, less invasive, and provides a lower complication rate during continuous IV administration. In addition, mini midline catheters can be left in place for 1-4 weeks, reducing the number of catheterizations. Mini-midline catheter placement sites include the forearm, anterior elbow fossa, or upper arm, and generally do not exceed the middle of the upper arm.20 The 2021 edition of the Infusion Therapy Standards of Practice (the "Standards") states that cephalic, vital, and median veins should be considered for placement of catheters, and that The standard indicates that the placement should be in the forearm, not exceeding the elbow socket, but the description is vague, and the level of evidence is Grade III. In addition to this, the domestic industry standards, the Technical Operation Code for Intravenous Therapy Nursing and related intravenous therapy guidelines do not provide clear standards and specifications for the use of mini-median catheters, and the selection of the optimal site is crucial to reducing complications.

Overseas studies have applied mini midline catheters to cardiac surgery and ICU patients, with the catheter placed in the upper arm, and the incidence of each complication is lower. In a study of mini midline catheter placement in children, the duration of retention was greater in the upper arm than in the forearm. Although several studies have reported differences in incidence and catheter retention time between the forearm and upper arm for mini midline catheters, few studies have directly compared the outcome of catheter placement in the upper arm or forearm, and there is very little direct experimental data on the relative advantages of the forearm versus the upper arm. Therefore, this study applies the mini midline catheter to patients and observes the application effect of different catheterization sites, aiming to provide a reference basis for patients to choose the optimal catheterization site, so as to reduce the occurrence of complications, prolong the catheter retention time, and alleviate the patient's pain.

ELIGIBILITY:
Inclusion Criteria:

* The expected duration of IV fluids before placement is 1-4 weeks.
* Intravenous fluids are used only during hospitalization.
* The nature of the infused drugs is in accordance with the indications for peripheral venous catheters.
* Conscious and able to communicate normally.
* Voluntarily participate in this study and sign the informed consent form.

Exclusion Criteria:

* History of radiation therapy, thrombosis, and trauma at the site of placement.
* Vulnerable groups, including those with mental illness, cognitive impairment, critically ill patients, pregnant women, illiterates, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Incidence of catheter-related complications | during catheter indwelling procedure
  Catheter-related complications included phlebitis, catheter-related thrombosis, catheter-related infection, catheter occlusion, catheter prolapse, blood leakage, and fluid leakage, and the incidence rate of each complication was the number of patients with the complication/total number of patients. The total incidence of catheter-related complications was the main outcome indicator, i.e., the number of patients with complications/the total number of patients, and the occurrence of one or more complications in the same patient was counted as one case.

CONTACTS AND LOCATIONS:
Overall Officials: Linfang Zhao, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Linfang Zhao, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cano A, Ettcheto M, Espina M, Lopez-Machado A, Cajal Y, Rabanal F, Sanchez-Lopez E, Camins A, Garcia ML, Souto EB. State-of-the-art polymeric nanoparticles as promising therapeutic tools against human bacterial infections. J Nanobiotechnology. 2020 Oct 31;18(1):156. doi: 10.1186/s12951-020-00714-2. PMID 33129333